CLINICAL TRIAL: NCT01413243
Title: Trichuris Suis Ova (TSO)in Recurrent Remittent Multiple Sclerosis and Clinically Isolated Syndrome - A Monocentric, Prospective, Randomized, Double-blind and Placebo-controlled Phase 2 Trial
Brief Title: Trichuris Suis Ova (TSO)in Recurrent Remittent Multiple Sclerosis and Clinically Isolated Syndrome
Acronym: TRIOMS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Berit Rosche, Dr. med., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TRIOMS-01
Record Dates: First submitted 2011-08-08; First posted 2011-08-10 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: Multiple Sclerosis
Keywords: Multipe sclerosis, Trichuris suis ova
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug: Trichuris suis ova (Experimental): Experimental: Trichuris suis ova (TSO) 2500 eggs every 2 weeks for 12 months
  Interventions: Drug: Trichuris suis ova
- Placebo (Placebo Comparator): Drug: Placebo, fluid every 2 weeks
  Interventions: Drug: Trichuris suis ova

INTERVENTIONS:
Drug: Trichuris suis ova — Trichuris suis ova 2500 eggs every 2 weeks
  Other Names: TSO

SUMMARY:
Trichuris suis ova (TSO) is a probiotic treatment based on the hygiene hypothesis, that has proven safe and effective in autoimmune inflammatory bowel disease. Clinical trails indicate that helminth infections have an immunomodulatory effect in multiple sclerosis as well. Investigators hypothesize that TSO® 2500 eggs given oral every 2 weeks for 12 months is - due to its immunomodulatory and antiinflammatory effect - in recurrent remittent multiple sclerosis and clinically isolated syndrome significantly more effective than an oral placebo treatment as assed by new T2 lesions in cerebral magnetic resonance imaging and clinical examination.

DETAILED DESCRIPTION:
TSO has an impact on the Th1-Th2 balance and effects Il-10 producing B-cells, mechanisms that result in an antiinflammatory effect.

A 12 month treatmet with TSO is safe and well-tolerated

ELIGIBILITY:
Inclusion Criteria:

* active Recurrent remittent Multiple Scleosis or Clinically isolated Syndrome
* inefficacy or intolerance for a therapy with Interferon-beta
* age 18 - 65
* EDSS <4

Exclusion Criteria:

* secondary or primary chronic progressive Multiple Sclerosis
* Immunomodulatoric or immunosuppressive therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-09; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Cumulative number of new T2 hyperintensive in cerebral magnetic resonance imaging (MRI) | after 12 months of treatment

SECONDARY OUTCOMES:
reduction NAA/Cr-ratio in MR-spectroscopy | after 12 month of treatment
Number of new Gadolinium lesions in magnetic resonance imaging (MRI) cerebral magnetic resonance imaging (MRI) | after 12 months of treatment
Volume of new T2 hyperintensive in cerebral magnetic resonance imaging (MRI) | after 12 months of treatment
Number of relapes, proression of diability measured in EDSS (Expanded Disability Status Scale) and MSFC (Multiple Sclerosis Functional Composite), | after 12 months of treatment
Number of Participants with Adverse Events | participants will be followed for the duration of the study and have every 3 month planed visits.

CONTACTS AND LOCATIONS:
Overall Officials: Berit Rosche, M.D., Principal Investigator — Charité-University; Friedemann Paul, M.D., Study Chair — Charité - University, NeuroCure Clinical Research Center
Locations (1):
- Charité - Universitätsmedizin Berlin, Department of Neurology, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Rosche B, Wernecke KD, Ohlraun S, Dorr JM, Paul F. Trichuris suis ova in relapsing-remitting multiple sclerosis and clinically isolated syndrome (TRIOMS): study protocol for a randomized controlled trial. Trials. 2013 Apr 25;14:112. doi: 10.1186/1745-6215-14-112. PMID 23782752